CLINICAL TRIAL: NCT06660901
Title: Cannabinoid Hyperemesis Syndrome. Prospective Multicenter Study of Patients Admitted to Adult Emergency Departments in Maine-et-Loire.
Acronym: CANN-AIE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC24_0175
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: D000096704; Cannabinoid Hyperemesis Syndrome
Keywords: marijuana; cannabis; Recurrent vomiting; nausea; abdominal pain; compulsive hot bathing behavior
MeSH Terms: conditions — Cannabinoid Hyperemesis Syndrome; Marijuana Abuse; Vomiting; Nausea; Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cannabinoid hyperemesis syndrome

SUMMARY:
Cannabinoid hyperemesis syndrome (CHS) is characterized by incoercible abdominal pain and vomiting in patients with chronic cannabis use. Patients are relieved by hot showers, an easily performed diagnostic test.

The prevalence of this syndrome in France is not well known. A single French study from 2021, carried out in two Marseille emergency departments, estimated a 1.6% prevalence of CHS (48 cases / 2848 patients) in patients consulting for acute abdominal pain with no etiology found over a 10-month period.

Cannabis is the most widely used illicit substance in France. France is also the second biggest cannabis consumer in Europe, with around 11% of the French population currently using the drug (use within the year).

Despite growing attention to CHS, the diagnosis and management of this syndrome remains difficult, with repeated visits to emergency departments often required before a diagnosis is made. What's more, once the diagnosis has been made, the severity of symptoms can lengthen the emergency room length of stay.

Main objective:

To estimate the incidence of cannabinoid hyperemesis syndrome among patients admitted on a first visit for abdominal pain and/or vomiting to the Maine et Loire emergency department.

Primary endpoint:

The incidence of cannabinoid hyperemesis syndrome among patients presenting with abdominal pain and/or vomiting, consulting adult emergency departments in Maine et Loire. Cannabinoid hyperemesis syndrome will be considered in all patients admitted for abdominal pain and/or vomiting, who are regular cannabis users (weekly use for more than 6 months declared by questionnaire) and in whom no other etiology is accepted after any additional examinations.

Research plan and procedure:

It is an observational, prospective, multi-center cohort study. Participation in the study is offered to any emergency room patient who meets all inclusion criteria and none of the non-inclusion criteria. Patients are included after reading the information note. Consent is obtained on a no-objection basis.

A questionnaire is given to participants via a QR code with an identification number generated by the investigating physician. This QR code opens an online questionnaire that the patient can fill in while in the emergency department. In the absence of access to the QR code (no cell phone), the questionnaire will be given to the participant in paper format by the investigating physician. It will be collected at the end of the inclusion visit.

Participants who have revealed cannabis use (at least 1 time per week for at least 6 months) via the questionnaire are followed up at 3 months (+/- 15 days) by telephone to assess the evolution of symptoms, any recurrences, medical treatment and whether or not cannabis has been withdrawn.

Inclusion criteria:

* Patients aged 18 to 65 years,
* Consulted an adult emergency department in Maine et Loire for abdominal pain and/or vomiting for the 1st time during the study period.

Non-inclusion criteria:

* Refusal to participate in the study
* Patient unable to answer the questionnaire (allophone, under guardianship, under protection, incapable of major age, in the process of legal proceedings)
* Pregnant women

Number of research participants:

At present, there are no data on the incidence of CHS in the French literature. In order to assess the number of subjects required, we made a projection based on the only French study to date. In this study, carried out in two departments in Marseille, the percentage of patients with CHS among those consulting the emergency department for acute abdominal pain was 1.6%. Thus, assuming that the proportion of the event will be identical to that of the study carried out in Marseille, i.e. 1.6%, it would be necessary to recruit 3,000 people with abdominal pain and/or vomiting to have around 50 patients with CHS.

Research duration:

Inclusion period: 12 months Duration of participation: 3 months +/- 15 days (for patients with CHS) Study duration: 15 months

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 65 years,
* Consulted the Maine et Loire adult emergency department for abdominal pain and/or vomiting for the 1st time during the study period.

Exclusion Criteria:

* Refusal to participate in the study
* Patient unable to answer questionnaire (allophone, under guardianship, under protection, incapable of age, under legal proceedings)
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: At present, there are no data on the incidence of CHS in the French literature. In order to assess the number of subjects required, we made a projection based on the only French study to date. In this study, carried out in two departments in Marseille, the percentage of patients with CHS among those consulting the emergency department for acute abdominal pain was 1.6%. Thus, assuming that the proportion of the event will be identical to that of the study carried out in Marseille, i.e. 1.6%, it would be necessary to recruit 3,000 people with abdominal pain and/or vomiting to have around 50 patients with CHS.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with confirmed cannabinoid hyperemesis syndrome (CHS) among patients presenting with abdominal pain and/or vomiting, consulting adult emergency departments in Maine et Loire | Inclusion period will last 12 month and the whole study 15 month. Participation of each CHS positive patient is expected to last 3 month +/- 15 days.
  The incidence of cannabinoid hyperemesis syndrome among patients presenting with abdominal pain and/or vomiting, consulting adult emergency departments in Maine et Loire. Cannabinoid hyperemesis syndrome will be considered in all patients admitted for abdominal pain and/or vomiting, who are regular cannabis users (weekly use for more than 6 months declared by questionnaire) and in whom no other etiology is accepted after further investigations.

SECONDARY OUTCOMES:
Gender and age distribution of patients with cannabinoid hyperhaemesis syndrome (CHS) | Inclusion period will last 12 months and the whole study 15 months. Participation of each CHS positive patient is expected to last 3 months +/- 15 days.
  Socio-demographic data for the CHS population: gender, age
Description and Distribution of CHS patients across clinical characteristics listing | Inclusion period will last 12 months and the whole study 15 months. Participation of each CHS positive patient is expected to last 3 months +/- 15 days.
  Clinical characteristics of patients with CHS:
  frequency, type and location of abdominal pain, schedule of vomiting, improved by hot shower or not.
Describe cannabis use in patients with CHS: duration and frequency of use | Inclusion period will last 12 months and the whole study 15 months. Participation of each CHS positive patient is expected to last 3 months +/- 15 days.
Describe hospital management and therapies used for patients with CHS: additional tests performed, effectiveness of therapies (analgesics, antiemetics), patient pathway (discharge, short-term hospitalization unit, hospitalization). | Inclusion period will last 12 months and the whole study 15 months. Participation of each CHS positive patient is expected to last 3 months +/- 15 days.
Number of cannabis withdrawal attempts at 3 months in patients with CHS | 3 months +/- 15 days
Number of patients with recurrence of symptoms (abdominal pain and/or vomiting) at 3 months | 3 monts +/- 15 days
Number of patients reporting total cessation of cannabis use at 3 months post-inclusion | 3 months +/- 15 days
Number of patients who need to consult again (emergency, general practitioner, other) at 3 months | 3 months +/- 15 days
Number of patients reporting a consultation with an addictology referral at 3 months | 3 months +/- 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Julien DENIS, Doctor, Principal Investigator — Saumur Hospital Center
Locations (3):
- France (3):
  - Angers Centre Hospitalier Universitaire (CHU), Angers
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier de Saumur, Saumur

IPD SHARING:
Plan to Share IPD: No